CLINICAL TRIAL: NCT00525135
Title: A Phase II Trial of Valproic Acid (Depakote ER ®) in Patients With Advanced Thyroid Cancers of Follicular Origin, Who Are Thyroglobulin Positive/RAI Unresponsive
Brief Title: Valproic Acid (Depakote ER) in Patients With Advanced Thyroid Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left university and study was halted prematurely. No data was analyzed.
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Valproic Acid
Record Dates: First submitted 2007-08-28; First posted 2007-09-05 (Estimated); Results first posted 2015-02-03 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-01

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): If a patient exhibits increased radioiodine uptake on the Thyrogen scan post valproic acid therapy, patients will then prepare for ablative treatment and will remain on valproic acid for a total of 16 weeks, until receiving RAI ablation.
  Interventions: Drug: Valproic Acid
- 2 (Other): If no increased uptake is seen, patients will continue on valproic acid for 6 additional weeks at an increased dosage, totaling an overall treatment time of 16 weeks as well.
  Interventions: Drug: Valproic Acid

INTERVENTIONS:
Drug: Valproic Acid — OUTLINE: This is a pilot study.
  Patients receive valproic acid daily for 16 weeks. Dose increases on Days 4 and 8; dose remains the same for weeks 2-10. All patients will undergo a Thyrogen® (thyrotropin alfa for injection) RAI scan at entry to the study and after completion of 10 weeks of valproic acid treatment.
  Quality of life is assessed at the end of every week through a study diary.
  Patients are followed at 1, 2, 4, 6, 8, 10, 12, 14, 16, and 17 (Schedule 1) weeks. Patients return for follow-up at 3, 6, and 12 months.

SUMMARY:
RATIONALE: Drugs such as valproic acid may make thyroid cancers more radioiodine sensitive, which will allow for detection of tumor and make further ablation treatment effective.

DETAILED DESCRIPTION:
PURPOSE: This phase II trial is studying how well valproic acid works in treating patients with thyroid cancers that do not respond well to other treatments.

ELIGIBILITY:
INCLUSION CRITERIA:

DISEASE CHARACTERISTICS

* Diagnosis of advanced/poorly differentiated thyroid cancer of follicular cell origin that is radioiodine-unresponsive
* Cumulative dose of radioiodine < 800 mCi
* No radioiodine uptake on whole body scan within 18 months of enrollment
* Inoperable extensive locoregional tumor mass and/or metastatic spread
* Failed conventional therapy that included total thyroidectomy AND radioactive iodine I 131 ablation
* Elevated thyroglobulin level (>2ng/ml on thyroid hormone, >10ng/ml off thyroid hormone)or Tg-antibody positive

PATIENT CHARACTERISTICS

-18 years or older

Entry lab results:

* Hemoglobin > 8.0 gm/dl
* Absolute Neutrophil Count > 750 cells/mm3
* Platelet count > 75000/mm3
* BUN < 1.5 times upper limit of normal (ULN)
* Creatinine < 1.5 times ULN
* Total protein > 6.4
* Total bilirubin should be < 1.5 times ULN.
* AST (SGOT), ALT (SGPT), ALKP and amylase < 1.5 times ULN
* Amylase < 1.5 times ULN
* Albumin > 2.5
* Ammonia < 1.5 times ULN

EXCLUSION CRITERIA:

* Not pregnant
* No nursing within the past 3 months
* No allergy to valproic acid
* No coexisting malignancy other than basal cell carcinoma
* No hepatic disease or significant dysfunction
* Karnofsky score > 80
* No pancreatitis
* No kidney dysfunction
* Fertile patients must use effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Electron Kebebew, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Comprehensive Cancer Center, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Intervention: Patients receive valproic acid daily for 16 weeks.
Period: Overall Study
Arm/Group | Study Intervention
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Intervention
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | NA (NA) — Due to a registration error, the PI did not receive notifications to report results until after the data retention period had passed; numeric data are no longer available for analysis.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Due to a registration error, the PI did not receive notifications to report results until after the data retention period had passed; numeric data are no longer available for analysis.
  Male | NA — Due to a registration error, the PI did not receive notifications to report results until after the data retention period had passed; numeric data are no longer available for analysis.
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Decrease in Thyroglobulin Level
Description: Number of participants with decreased thyroglobulin level after study treatment
Time Frame: Baseline, 16 weeks
Measure: Number; unit: participants
Arm/Group | Study Intervention
Number analyzed (Participants) | 5
participants | 0

2. Secondary Outcome: Increased Radioactive Iodine Uptake
Description: Number of participants with increased radioiodine uptake on the Thyrogen scan post valproic acid therapy
Time Frame: Baseline, 10 weeks
Measure: Number; unit: participants
Arm/Group | Study Intervention
Number analyzed (Participants) | 5
participants | 3

3. Secondary Outcome: Side Effects of Drugs Affecting Quality of Life
Description: Number of participants experiencing > Grade 1 adverse events (including fatigue) attributable to study treatment
Time Frame: 17 weeks
Measure: Number; unit: participants
Arm/Group | Study Intervention
Number analyzed (Participants) | 5
participants | 0

4. Primary Outcome: Decrease in Tumor Size
Description: Number of participants with decreased tumor size after study treatment
Time Frame: Baseline, 16 weeks
Measure: Number; unit: participants
Arm/Group | Study Intervention
Number analyzed (Participants) | 5
participants | 0

5. Secondary Outcome: Survival
Time Frame: up to 10 years post-study treatment
Population: Due to early termination, participants were not followed for survival after the primary outcome timeframe
Arm/Group | Study Intervention
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 17 weeks
Arm/Group | Study Intervention
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes